CLINICAL TRIAL: NCT01469689
Title: Raising Awareness of Online Therapies for Depression: Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Plymouth (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Principal Investigator, Ray Jones, Professor of Health Informatics, University of Plymouth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RR103348-101
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Depression
Keywords: People; living; community
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Google Adwords only (Experimental): In these areas,the investigators will display online adverts using Google Adwords, with links to the investigators' project website, and from there to four other websites for depression.
  Interventions: Other: Google Adwords
- Local organisation websites (Experimental): In these areas, the investigators will try to place adverts on the websites of local organizations, with links to the investigators' project website, and from there to four other websites for depression.
  Interventions: Other: Local organisation websites
- Google Ads and local websites (Experimental): In these areas, the investigators will place Google Adwords and also try to place adverts on the websites of local organizations, with links to the investigators' project website, and from there to four other websites for depression.
  Interventions: Other: Google Adwords; Other: Local organisation websites
- Control (No Intervention): Control areas. No Intervention

INTERVENTIONS:
Other: Google Adwords — The investigators will display Google Adwords advertising the investigators' website offering online help for depression
  Arms: Google Ads and local websites; Google Adwords only
Other: Local organisation websites — The investigators will place adverts on local organization websites with links to the investigators' project website offering online help for depression
  Arms: Google Ads and local websites; Local organisation websites

SUMMARY:
Web based cognitive behavioural therapy (webCBT) for depression is recommended by NICE but analysis of the geographic distribution of one webCBT site showed 15-fold variation in use across Britain. Such variation is unlikely to be from differences in prevalence. Raising awareness of webCBT could benefit many people with depression but it is not clear how direct-to-patient promotion online or via the media, compares with GP centred methods. This pilot cluster randomised controlled trial will explore the use of online methods to raise awareness in preparation for subsequent study comparing different approaches.

In a pilot cluster randomised trial the investigators will explore the feasibility and likely impact of online methods of raising awareness of webCBT, assessing how many people with depression respond to geographically restricted Google and local website advertisements. The investigators will explore costs of recruitment and define and document the best online methods that might subsequently be used in a definitive trial comparing online with mass media and GP centred methods for raising awareness. The investigators will compare intervention with control areas to estimate impact on registration levels and compare rate of completion of webCBT of these 'additional' registrants with other registrants. Recommendations will be made for a subsequent trial comparing online with other methods.

ELIGIBILITY:
Inclusion Criteria:

* people living in Britain searching for online help for depression

Exclusion Criteria:

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8231 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Registration on Living Life To The Full website | 9 months
  This is a cluster trial with primary outcome the number of registrations for given geographical areas on a website (Living Life to The Full) offering cognitive behaviuoural therapy for depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Online, Plymouth, United Kingdom

REFERENCES:
- [Derived] Jones RB, Goldsmith L, Hewson P, Williams CJ. Recruitment to online therapies for depression: pilot cluster randomized controlled trial. J Med Internet Res. 2013 Mar 5;15(3):e45. doi: 10.2196/jmir.2367. PMID 23462072
- [Derived] Jones RB, Goldsmith L, Williams CJ, Kamel Boulos MN. Accuracy of geographically targeted internet advertisements on Google AdWords for recruitment in a randomized trial. J Med Internet Res. 2012 Jun 20;14(3):e84. doi: 10.2196/jmir.1991. PMID 22718043
- [Derived] Jones RB, Goldsmith L, Hewson P, Kamel Boulos MN, Williams CJ. Do adverts increase the probability of finding online cognitive behavioural therapy for depression? Cross-sectional study. BMJ Open. 2012 Apr 16;2(2):e000800. doi: 10.1136/bmjopen-2011-000800. Print 2012. PMID 22508957
- See also: University of Plymouth (Sponsoring organisation) — http://www.plymouth.ac.uk
- See also: Collaborating centre — http://www.glasgow.ac.uk